CLINICAL TRIAL: NCT05899946
Title: An Integrated Program Led by Nursing Students as Peer Role Models With Robots to Promote Anti-cannabis Messages in Parents and Their Children
Brief Title: An Integrated Program to Promote Anti-cannabis Messages
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Katherine Lam, Research Assistant Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Anti-cannabis promoting
Record Dates: First submitted 2023-05-11; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Cannabis
Keywords: Nursing Students; Child; Parents
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pre- and post-educational group (Other): This project will deliver an integrated program by nursing students with robots to clarify the misunderstanding about cannabis among parents and their children in Hong Kong
  Interventions: Other: A community-based network training program

INTERVENTIONS:
Other: A community-based network training program — A 3-phase program including establishing a community-based network, video competition, and Video promotions will be conducted.

SUMMARY:
The number of youngsters abusing cannabis is surging, the public health consequences caused by cannabis can be unpredictable. Educating the public especially the young population about cannabis need to be highlighted. To successfully promote anti-cannabis messages to youngsters and prevent them from taking cannabis, the involvement of their parents and modern technology such as robots can be helpful. This project aims to educate the young population and their parents about cannabis, particularly its legal consequences and clarifying their misconceptions.

DETAILED DESCRIPTION:
A pre-post study design will be used. A total of 50 nursing students and 150 parent-child-dyads will be recruited by sending mass emails or sending invitation letters. The nursing students are in their year 2 or above bachelor program in the Hong Kong Polytechnic University. The inclusion criteria for parent-child-dyads include: (1) children who are aged 13 - 20, (2) children who have a parent who are willing to join with the child, and (3) parent-child dyads who are able to speak in Cantonese and write in Chinese. The outcome measures will cover demographic data, the knowledge about cannabis-related harm, the permissive attitude towards smoking cannabis and drugs trafficking.

ELIGIBILITY:
Inclusion Criteria

* children who are aged 13 - 20
* children who have a parent who are willing to join with the child

Exclusion Criteria:

-parents and children who are not able to speak Cantonese and write in Chinese

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The Beat Drugs Fund Question Set No. 24 for knowledge at baseline | at baseline
  The Beat Drugs Fund Question Set No. 24 (Knowledge about Cannabis-related Harms Pre/post-activity Evaluation Questionnaire) will be used to measure the knowledge about cannabis-related harm among youngsters and their parents, and the nursing students
The Beat Drugs Fund Question Set No. 24 for knowledge at the end of educational workshops completion | at the end of educational workshops completion, an average of 10 months
  The Beat Drugs Fund Question Set No. 24 (Knowledge about Cannabis-related Harms Pre/post-activity Evaluation Questionnaire) will be used to measure the knowledge about cannabis-related harm among youngsters and their parents, and the nursing students
The BDF Question Set No. 25 for attitude towards Smoking Cannabis at baseline | at baseline
  The BDF Question Set No. 25 (Permissive Attitude towards Smoking Cannabis Pre/Post-Activity Evaluation Questionnaire) will be used to assess the permissive attitude towards smoking cannabis among youngsters and their parents, and the nursing students
The BDF Question Set No. 25 for attitude towards Smoking Cannabis at the end of educational workshops completion | at the end of educational workshops completion, an average of 10 months
  The BDF Question Set No. 25 (Permissive Attitude towards Smoking Cannabis Pre/Post-Activity Evaluation Questionnaire) will be used to assess the permissive attitude towards smoking cannabis among youngsters and their parents, and the nursing students
The BDF Question Set No. 26 for attitude towards drugs trafficking at baseline | at baseline
  The BDF Question Set No. 26 (Questionnaire to Measure Attitude towards Drug Trafficking) will be used to record the permissive attitude towards drugs trafficking among youngsters and their parents, and the nursing students
The BDF Question Set No. 26 for attitude towards drugs trafficking at the end of educational workshops completion | at the end of educational workshops completion, an average of 10 months
  The BDF Question Set No. 26 (Questionnaire to Measure Attitude towards Drug Trafficking) will be used to record the permissive attitude towards drugs trafficking among youngsters and their parents, and the nursing students

CONTACTS AND LOCATIONS:
Overall Officials: Ka Wai Katherine Lam, Principal Investigator — School of Nursing, Hong Kong Polytechnic University
Locations (1):
- Katherine Lam, Hong Kong, Hong Kong,China, Hong Kong

IPD SHARING:
Plan to Share IPD: No